CLINICAL TRIAL: NCT05682989
Title: Evaluation of Efficacy and Safety of Urogynecology Synthetic Mesh Surgery in Women With Pelvic Organ Prolapse
Brief Title: Efficacy/Safety of Urogynecology Synthetic Mesh Surgery
Status: Recruiting | Type: Observational
Sponsor: Mackay Medical College (Other)
Responsible Party: Principal Investigator, Chin-Tsung Shen, The Office of Research and Development, Mackay Medical College
Other Study IDs: 22MMHIS361e
Record Dates: First submitted 2022-12-28; First posted 2023-01-12 (Actual); Last update posted 2023-04-05 (Actual); Status verified 2023-04

CONDITIONS: Pelvic Organ Prolapse; Stage III and IV High Grade Pelvic Organ Prolapse
MeSH Terms: conditions — Pelvic Organ Prolapse

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- mesh surgery: Data obtained before the operation
  Interventions: Procedure: Urodynamic investigations before and after a mesh surgery protocol.
- Robotic-assisted sacrocolpopexy: Data obtained before the operation
  Interventions: Procedure: Urodynamic investigations before and after a robotic-assisted sacrocolpopexy protocol.
- a hysterectomy with trans-vaginal mesh repair (Surelift®, Neomedic International, Barcelona, Spain): Data obtained before the operation
  Interventions: Procedure: Urodynamic investigations before and after a hysterectomy with trans-vaginal mesh repair

INTERVENTIONS:
Procedure: Urodynamic investigations before and after a mesh surgery protocol. — Urodynamic investigations (The urodynamic study included free uroflowmetry, postvoid residual, filling and voiding cystometry, and a urethral pressure profile. The filling cystometry and urethral pressure profile were performed with 37 degrees C normal saline similar to body temperature at an infusion rate of 80 ml/min.
  Groups: mesh surgery
Procedure: Urodynamic investigations before and after a robotic-assisted sacrocolpopexy protocol. — All surgeries were performed using a DaVinci robotic system (Intuitive® Surgical Inc., Sunnyvale, California,US) with standardized technique and materials. Patients were positioned in dorsal lithotomy and steep Trendelenburg position. Trocars were placed bilaterally, and an assistant port was placed laterally. The peritoneum was opened medial to the ureter to develop an avascular space. The mesh was placed on the posterior and anterior vaginal wall and fixed at the level of anterior longitudinal ligaments S1/S2 by sutures. An intraoperative clinical examination was performed to ensure the mesh was in a tension-free position.
  Groups: Robotic-assisted sacrocolpopexy
Procedure: Urodynamic investigations before and after a hysterectomy with trans-vaginal mesh repair — In summary, a vertical incision was made in the anterior vaginal wall to access the vesicovaginal space. The sacrospinous ligament was dissected, and an applicator was inserted and positioned over the SSL. The anchor was fixed to the SSL and the thread was attached to the mesh. The mesh was then adjusted in a tension-free manner, excess mesh was cut, and the incision was closed with suture.
  Groups: a hysterectomy with trans-vaginal mesh repair (Surelift®, Neomedic International, Barcelona, Spain)

SUMMARY:
This is a retrospective cohort study, aiming at analyzing the efficacy and safety of mesh surgery in pelvic organ prolapse. The synthetic mesh for pelvic organ prolapse include transvaginal mesh or laparotomy, laparoscope, or robotic-assisted laparoscopic sacrocolpopexy with mesh augmentation. The investigators would like to evaluate the efficacy and safety, such as recurrence rates and complication rates for women who underwent urogynecology mesh surgery.

DETAILED DESCRIPTION:
Gynecologic mesh, including transvaginal mesh and mesh used in abdominal or laparoscopic sacrocolpopexy, has been used for pelvic organ prolapse since its debut in the US in 2005. It provides higher success and satisfaction rate than traditional colporrhaphy, but mesh-related complications, such as pain, mesh exposure and bleeding, have been reported. U.S. Food and Drug Administration issued a Safety Update in 2011 to inform the public that serious complications associated with synthetic mesh for the transvaginal repair of POP were common. Taiwan FDA and associated committees decided that the use of gynecologic mesh should be regulated. Thorough study and evaluation are needed.

ELIGIBILITY:
Inclusion Criteria:

* Pelvic organ prolapse patients with objective / subjective voiding dysfunctions
* Underwent surgery for symptomatic POP ≥ stage II (POP-Q system)

Exclusion Criteria:

* Patients with a history of pelvic radiation.
* Patients with a history of vesico-/recto-/urethra-vaginal fistula
* Patients unable to be followed up.

Ages: 30 Years to 100 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: History of POP patients with concurrent objective and/or subjective voiding dysfunctions who underwent primary TVM surgery for symptomatic POP
  ≥ stage II (POP Quantification system; POP-Q system) in Mackay Memorial Hospital were recruited.
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2023-08-01 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
trans-vaginal mesh repair | Generally in our hospital, pre-operative investigation will be done about 30 days before surgery, post-operative investigation will within 1year after surgery.
  Urodynamic investigations (The urodynamic study included free uroflowmetry, postvoid residual, filling and voiding cystometry, and a urethral pressure profile. The filling cystometry and urethral pressure profile were performed with 37 degrees C normal saline similar to body temperature at an infusion rate of 80 ml/min.
  1. The urodynamic data of POP patient with grade > or = II, will be retrograde analyzed and and compared.
  2. Pressure-associated parameters, such as abdominal pressure (Pabd), detrusor pressure (Pdet) will be measured as centimeter of water column (cmH2O), volume-associated parameters, such as infused volume (Vinf), voided volume (Vvod) and intravesical volume (Vive) will measured as ml. Derived parameter will be expressed as their results of calculation.

CONTACTS AND LOCATIONS:
Overall Officials: Hui-Hsuan Lau, M.D., Study Chair — Department of Ear, Nose, and Throat, MacKay Memorial Hospital, Taipei, Taiwan
Locations (1):
- Department of Obstetrics and Gynecology, New Taipei City, Taiwan

IPD SHARING:
Plan to Share IPD: No
For we uncertain if this might violate personal information laws in our country.

REFERENCES:
- [Background] Abrams P, Andersson KE, Birder L, Brubaker L, Cardozo L, Chapple C, Cottenden A, Davila W, de Ridder D, Dmochowski R, Drake M, Dubeau C, Fry C, Hanno P, Smith JH, Herschorn S, Hosker G, Kelleher C, Koelbl H, Khoury S, Madoff R, Milsom I, Moore K, Newman D, Nitti V, Norton C, Nygaard I, Payne C, Smith A, Staskin D, Tekgul S, Thuroff J, Tubaro A, Vodusek D, Wein A, Wyndaele JJ; Members of Committees; Fourth International Consultation on Incontinence. Fourth International Consultation on Incontinence Recommendations of the International Scientific Committee: Evaluation and treatment of urinary incontinence, pelvic organ prolapse, and fecal incontinence. Neurourol Urodyn. 2010;29(1):213-40. doi: 10.1002/nau.20870. No abstract available. PMID 20025020
- [Background] GREEN TH Jr. Development of a plan for the diagnosis and treatment of urinary stress incontinence. Am J Obstet Gynecol. 1962 Mar 1;83:632-48. doi: 10.1016/s0002-9378(16)35894-x. No abstract available. PMID 13901453
- [Background] McGuire EJ, Lytton B, Kohorn EI, Pepe V. The value of urodynamic testing in stress urinary incontinence. J Urol. 1980 Aug;124(2):256-8. doi: 10.1016/s0022-5347(17)55396-3. PMID 7401242
- [Background] Ulmsten U, Johnson P, Rezapour M. A three-year follow up of tension free vaginal tape for surgical treatment of female stress urinary incontinence. Br J Obstet Gynaecol. 1999 Apr;106(4):345-50. doi: 10.1111/j.1471-0528.1999.tb08272.x. PMID 10426241
- [Background] Fusco F, Abdel-Fattah M, Chapple CR, Creta M, La Falce S, Waltregny D, Novara G. Updated Systematic Review and Meta-analysis of the Comparative Data on Colposuspensions, Pubovaginal Slings, and Midurethral Tapes in the Surgical Treatment of Female Stress Urinary Incontinence. Eur Urol. 2017 Oct;72(4):567-591. doi: 10.1016/j.eururo.2017.04.026. Epub 2017 May 4. PMID 28479203
- [Background] Jiao B, Lai S, Xu X, Zhang M, Diao T, Zhang G. A systematic review and meta-analysis of single-incision mini-slings (MiniArc) versus transobturator mid-urethral slings in surgical management of female stress urinary incontinence. Medicine (Baltimore). 2018 Apr;97(14):e0283. doi: 10.1097/MD.0000000000010283. PMID 29620645
- [Background] Stav K, Dwyer PL, Rosamilia A, Schierlitz L, Lim YN, Lee J. Risk factors of treatment failure of midurethral sling procedures for women with urinary stress incontinence. Int Urogynecol J. 2010 Feb;21(2):149-55. doi: 10.1007/s00192-009-1020-9. Epub 2009 Oct 24. PMID 19855914
- [Background] Ford AA, Ogah JA. Retropubic or transobturator mid-urethral slings for intrinsic sphincter deficiency-related stress urinary incontinence in women: a systematic review and meta-analysis. Int Urogynecol J. 2016 Jan;27(1):19-28. doi: 10.1007/s00192-015-2797-3. Epub 2015 Jul 29. PMID 26220506
- [Background] Sand PK, Bowen LW, Panganiban R, Ostergard DR. The low pressure urethra as a factor in failed retropubic urethropexy. Obstet Gynecol. 1987 Mar;69(3 Pt 1):399-402. PMID 3822288
- [Background] McGuire EJ, Fitzpatrick CC, Wan J, Bloom D, Sanvordenker J, Ritchey M, Gormley EA. Clinical assessment of urethral sphincter function. J Urol. 1993 Nov;150(5 Pt 1):1452-4. doi: 10.1016/s0022-5347(17)35806-8. PMID 8411422
- [Background] Uebersax JS, Wyman JF, Shumaker SA, McClish DK, Fantl JA. Short forms to assess life quality and symptom distress for urinary incontinence in women: the Incontinence Impact Questionnaire and the Urogenital Distress Inventory. Continence Program for Women Research Group. Neurourol Urodyn. 1995;14(2):131-9. doi: 10.1002/nau.1930140206. PMID 7780440
- [Background] Kenton K, Stoddard AM, Zyczynski H, Albo M, Rickey L, Norton P, Wai C, Kraus SR, Sirls LT, Kusek JW, Litman HJ, Chang RP, Richter HE. 5-year longitudinal followup after retropubic and transobturator mid urethral slings. J Urol. 2015 Jan;193(1):203-10. doi: 10.1016/j.juro.2014.08.089. Epub 2014 Aug 23. PMID 25158274
- [Background] Foss Hansen M, Lose G, Kesmodel US, Gradel KO. Reoperation for urinary incontinence: a nationwide cohort study, 1998-2007. Am J Obstet Gynecol. 2016 Feb;214(2):263.e1-263.e8. doi: 10.1016/j.ajog.2015.08.069. Epub 2015 Sep 5. PMID 26344752
- [Background] Sun MJ, Chuang YL, Lau HH, Lo TS, Su TH. The efficacy and complications of using transvaginal mesh to treat pelvic organ prolapse in Taiwan: A 10-year review. Taiwan J Obstet Gynecol. 2021 Mar;60(2):187-192. doi: 10.1016/j.tjog.2021.01.031. PMID 33678316
- [Derived] Lau HH, Lai CY, Hsieh MC, Peng HY, Chou D, Su TH, Lee JJ, Lin TB. Uneven effects of trans-vaginal mesh reconstruction on the viscoelastic property of the urinary bladder in patients with pelvic organ prolapse. Front Bioeng Biotechnol. 2026 Jan 12;13:1677779. doi: 10.3389/fbioe.2025.1677779. eCollection 2025. PMID 41602457
- [Derived] Lau HH, Lai CY, Hsieh MC, Peng HY, Chou D, Su TH, Lee JJ, Lin TB. Pressure-volume analysis of thermodynamic workload of voiding - an application in pelvic organ prolapse patients subjected to robotic-assisted sacrocolpopexy. Biomed Eng Lett. 2024 Dec 30;15(2):357-365. doi: 10.1007/s13534-024-00453-5. eCollection 2025 Mar. PMID 40026886